CLINICAL TRIAL: NCT06337435
Title: The Ability of the Multi-Looped Lingual Retainer Activated by A New Method to Align Lower Incisor Crowding
Brief Title: Using Multi-looped Lingual Retainer to Relief Anterior Mandibular Crowding
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basel Mouafak Mohamed Alhawash, master degree faculty Cairo university, Cairo University
Other Study IDs: 8223
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: multi-looped wire — using multi-looped wire as a retainer

SUMMARY:
this study aim to evaluate the multi-looped lingual retainer activated by a new method to relief the anterior crowding

DETAILED DESCRIPTION:
1. patients preparation( photo- impression- x-ray- scan the lower cast to calculate the crowding )
2. The multi-looped lingual retainer was fabricated on the patient's lower cast
3. The lingual surfaces of teeth were etched with 35% phosphoric acid for 20 seconds The multi-looped lingual retainer was activated in the new way (Kattan method ) by tightening a steel ligature wire 0.010 inches, to the reinforcement 0.020-inch stainless steel arch-wire.
4. the bonding agent was applied on such surfaces after a good isolation and was light-cured for 20 seconds.
5. A flowable composite resin was applied. After checking its fit on the surface of the teeth, The lingual wire was bonded with a drop of flowable composite resin and was light-cured for 20 seconds.
6. follow-up the patients * Outcomes: The improvement of lower incisors irregularity using Little Irregularity Index.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, the ages of 16 to 25, the patients having class I canine with mild to moderate lower incisors crowding
* good oral hygiene.

Exclusion Criteria:

* Facial trauma, Oral habits such as onychophagia, pen biting, and tooth mobility.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with mild to moderate crowding
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
The improvement of lower incisors irregularity using Little Irregularity Index. | follow-up three to six months
  using multi-looped for relief crowding, the digital model analysis will be used to calculate the amount of irregularity by using Little Irregularity Index .the measurement will be done on 3-shape software.

SECONDARY OUTCOMES:
The stability of lower incisor positioning after ending treatment | after 1-3 months
  using multi-looped as a retainer for stability to prevent the relapse after end treatment and the amount of lower incisor irregularity will be evaluated on scanned post-treatment digital models and measured on the 3-shape software.

CONTACTS AND LOCATIONS:
Overall Officials: bassel mouafak alhawash, master, Principal Investigator — bassel.alhawash@dentistry.cu.edu.eg
Locations (1):
- faculty of dentistry Cairo university, Cairo, Egypt